CLINICAL TRIAL: NCT07179081
Title: Phase I Clinical Study on Dose-Escalation Tolerability and Pharmacokinetics of AL58805 in Patients With Advanced Tumors
Brief Title: A Study of AL58805 in Patients With Advanced Tumors
Status: Recruiting | Phase: Phase 1 | Type: Interventional
Sponsor: Advenchen Laboratories Nanjing Ltd. (Industry)
Responsible Party: Sponsor
Organization: Advenchen Laboratories, LLC (Industry)
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Screening
Other Study IDs: AL58805-CN-001B
Record Dates: First submitted 2025-09-05; First posted 2025-09-17 (Actual); Last update posted 2025-09-17 (Actual); Status verified 2025-09

CONDITIONS: Advanced Tumors

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- AL58805 (Experimental): 20mg 、40mg QD; 20mg 、30mg、40mg、50mg、60mg BID；
  Interventions: Drug: AL58805

INTERVENTIONS:
Drug: AL58805 — Oral,Multiple administrations, once or twice daily（20mg 、40mg QD; 20mg 、30mg、40mg、50mg、60mg BID；）

SUMMARY:
This Phase I clinical trial is a dose-escalation, multicenter study in patients with advanced solid tumors. It includes tolerance studies of sequential multiple oral doses of AL58805 and pharmacokinetic studies of single and multiple doses, analyzing the tolerance range of multiple doses, observing the maximum tolerated dose (MTD) and dose-limiting toxicity (DLT) in solid tumor patients, and assessing the reversibility of toxicity and the relationship between toxicity and dose.

ELIGIBILITY:
Inclusion Criteria:

Subjects must meet all the following criteria to be eligible:

1. Patients with histologically or cytologically confirmed advanced tumors (including but not limited to lymphoma, colorectal cancer, breast cancer, pancreatic cancer, lung cancer, head and neck cancer, bladder cancer, cholangiocarcinoma) who lack effective standard treatment options or have failed conventional standard treatments (due to disease progression or intolerable toxicity).
2. Previous treatment with cytotoxic chemotherapy, with at least 4 weeks between the end of chemotherapy and enrollment, and recovery from previous chemotherapy toxicities to ≤ Grade 1 (except alopecia).
3. Must have measurable lesions according to RECIST 1.1 criteria.
4. Major organ function: Absolute neutrophil count (ANC) ≥1.5 × 10^9/L (1500/mm3), platelets ≥75 × 10^9/L, hemoglobin ≥9g/dL. Serum total bilirubin ≤2 × upper limit of normal (ULN). Serum creatinine ≤1.5 × ULN or creatinine clearance ≥50 mL/min. For patients without liver metastases, alanine aminotransferase (ALT) and aspartate aminotransferase (AST) ≤2.5 × ULN; for patients with liver metastases, ALT and AST ≤5 × ULN. Left ventricular ejection fraction (LVEF) ≥ lower limit of normal.
5. Age ≥18 years; ECOG performance status (PS) 0 or 1.
6. Expected survival time of at least 12 weeks.
7. No malabsorption or other gastrointestinal diseases affecting drug absorption.
8. For women of childbearing potential: Negative pregnancy test before treatment and use of medically approved contraception during treatment and for 3 months after treatment ends. Must be non-lactating.
9. For male subjects: Surgical sterilization or use of medically approved contraception during treatment and for 3 months after treatment ends.

Ability to understand and sign informed consent.

Exclusion Criteria:

Subjects meeting any of the following criteria will be excluded:

1. Known allergy to the investigational drug or drugs with similar chemical structures.
2. Use of unapproved drugs or other investigational drugs within 30 days before enrollment.
3. Status of the organ systems:

   Current symptomatic brain metastases or leptomeningeal metastases, or central nervous system (CNS) metastases with uncontrolled symptoms within 8 weeks of first dose.

   Uncontrolled hypertension requiring multiple medications (Grade 2 or higher). Acute myocardial infarction within 6 months. Current arrhythmias (e.g., long QT syndrome, Bazett's corrected QTc ≥480 ms). NYHA Class III or IV heart failure. Poorly controlled diabetes. Any unstable systemic disease (including active infection, angina, hepatic, renal, or metabolic diseases).

   Presence of ascites or pleural effusion (CTCAE 5.0 ≥ Grade 2). Persistent diarrhea (average watery stools ≥1 per day). History of definite neurological or psychiatric disorders (e.g., epilepsy, dementia, mood disorders).
4. The functional level of each organ： Urine protein ≥++ and 24-hour urine protein >1.0 g. Patients treated with anticoagulants or vitamin K antagonists, such as warfarin, heparin, or their analogs, should have an international normalized ratio (INR) of prothrombin time ≤1.5. In this case, low-dose warfarin (1mg, orally, once daily) or low-dose aspirin (daily dose not exceeding 100mg) can be used for prophylactic purposes. All other conditions are considered exclusion criteria.

   Patients with active/venous thrombosis events within 6 months, such as cerebrovascular accidents (including transient ischemic attacks), deep vein thrombosis and pulmonary embolism.
5. Previous treatment with the investigational drug.
6. Patients exhibiting hepatitis B surface antigen (HBsAg) positivity with HBV DNA concentrations ≥10⁴ copies/mL (equivalent to 2000 IU/mL) must initiate antiviral therapy prior to study consideration. Eligibility for enrollment is contingent upon achieving sustained HBV-DNA suppression below these threshold values. Antiviral therapy will be maintained throughout the study period with concurrent monitoring of hepatic function parameters and quantitative HBV DNA levels. The exclusion criteria further encompass individuals with detectable HCV antibodies or HCV RNA, HIV seropositivity, congenital/acquired immunodeficiencies, or prior organ transplantation history.
7. Concurrent other anti-tumor treatments. Other conditions deemed unsuitable by the investigator.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 40 (Estimated)
Dates: Start 2020-12-20 (Actual); Primary Completion 2026-01-26 (Estimated); Study Completion 2026-01-26 (Estimated)

PRIMARY OUTCOMES:
Dose-limiting toxicity | From signing the ICF until 28 days after the first dosing
  It is the evaluation of dose-limiting toxicity (DLT) and general safety that occur during the single administration and the first continuous administration treatment cycle. The evaluation depends on the criteria for DLT. The parameters used to assess safety in this study include adverse events, physical examinations, vital signs (especially blood pressure), and laboratory tests (including serum chemistry, hematology, urine routine, and electrocardiogram (ECG), etc.)

SECONDARY OUTCOMES:
Tmax | Conduct testing within 1 month after all subjects collect plasma samples at all time points required by the protocol.
  Determine the time to reach maximum plasma concentration (Tmax) of AL58805 after single administration and continuous administration for 28 days.
Css_min | Conduct testing within 1 month after all subjects collect plasma samples at all time points required by the protocol.
  Measure the minimum steady - state plasma concentration (Css_min) of AL58805 during continuous administration for 28 days.
Css_av | Conduct testing within 1 month after all subjects collect plasma samples at all time points required by the protocol.
  Calculate the average steady - state plasma concentration (Css_av) of AL58805 during continuous administration for 28 days.
T1/2 | Conduct testing within 1 month after all subjects collect plasma samples at all time points required by the protocol.
  Estimate the elimination half - life (T1/2) of AL58805 after single administration and continuous administration for 28 days.
CL or CL/F | Conduct testing within 1 month after all subjects collect plasma samples at all time points required by the protocol.
  Assess the clearance (CL) or apparent clearance (CL/F) of AL58805 after single administration and continuous administration for 28 days.
AUCss | Conduct testing within 1 month after all subjects collect plasma samples at all time points required by the protocol.
  Evaluate the area under the steady - state plasma concentration - time curve (AUCss) of AL58805 during continuous administration for 28 days.
DF | Conduct testing within 1 month after all subjects collect plasma samples at all time points required by the protocol.
  Calculate the fluctuation index (DF) of AL58805 during continuous administration for 28 days.

CONTACTS AND LOCATIONS:
Overall Officials: Dongfang Li, Principal Investigator — Hunan Cancer Hospital; Yongchang Zhang, Principal Investigator — Hunan Cancer Hospital
Locations (1):
- Hunan Cancer Hospital, Changsha, Hunan, China

IPD SHARING:
Plan to Share IPD: No